CLINICAL TRIAL: NCT04054674
Title: Clinical Performance Of Lithium Disilicate Crowns Restoring Endodontically Treated Teeth With Two Occlusal Preparation Schemes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Salem, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBC-CU-2019920
Record Dates: First submitted 2019-08-07; First posted 2019-08-13 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Fracture of Lithium Disilicate (e.Max) Crowns
Keywords: e.max; occlusal scheme; endodontically treated teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- flat occlusal scheme restored by lithium disilicate crown (Experimental): flat occlusal preparation of endodontically treated teeth is performed clinically and then the final restorations will be lithium disilicate (e.max) crowns.
  Interventions: Procedure: Abutments with flat occlusal scheme preparation restored by lithium disilicate crowns
- planar occlusal scheme restored by lithium disilcate crown (No Intervention): planar occlusal preparation of endodontically treated teeth is performed clinically and then the final restorations will be lithium disilicate (e.max) crowns.

INTERVENTIONS:
Procedure: Abutments with flat occlusal scheme preparation restored by lithium disilicate crowns — Clinical trials lacks information about flat occlusal preparation design in case of endodontically treated teeth. Therefore, this is tested during preparation when compared to planer occlusal preparation while the final restoration in both arms is lithium disilicate (e.max) crowns.
  Arms: flat occlusal scheme restored by lithium disilicate crown

SUMMARY:
The aim of this study is to evaluate the clinical performance of lithium disilicate crowns restoring endodontically treated teeth with two occlusal preparation schemes.

DETAILED DESCRIPTION:
Statement of the problem:

The endodontically treated teeth need to be restored back to form, function and aesthetics. The quality of the coronal restoration will directly impact on their survival and success. The aim of the coronal restoration of endodontically treated teeth is to provide the necessary strength for the restoration/tooth complex through tooth preparation in order to withstand functional stress and prevent crown and/or root fracture. The use of ceramic crowns has increased substantially in recent years because of their superior esthetics and high mechanical properties. Long term success of all ceramic crowns is affected by many factors and the failure patterns of these all ceramic crowns should be inspected closely to detect their clinical performance.

Rationale for carrying out the trial:

Endodontic treatment weakens posterior teeth and ought to be covered by crowns.The capability of these crowns to bear load relies on the preparation of an appropriate design and the selection of a crown material with adequate fracture strength and thickness. In vital teeth, the anatomic occlusal preparation design is followed such that the occlusal surface is reduced uniformly, maintaining the cusps and normal inclined planes but at a reduced height. This aids in minimizing the risk of pulp injury. In contrast, in non-vital teeth, this design can be modified such that the occlusal surface is prepared in two planes (buccal and lingual planes). A flat prepared occlusal surface provides less quantitative and better qualitative stresses when compared to an anatomically prepared surface

ELIGIBILITY:
Inclusion Criteria:

* Have no active periodontal diseases or periapical pathosis
* No tooth mobility or furcation involvement with sufficient occluso-gingival height
* Psychologically and physically able to withstand conventional dental procedures
* Patients with good endodontically treated teeth indicated for full coverage restorations
* Able to return for follow-up examination and evaluation

Exclusion Criteria:

* Patient with active resistant periodontal diseases
* Patients with poor oral hygiene and uncooperative
* Pregnant women that won't be able to come for follow-up visits
* Patients in the growth stage with partially erupted teeth
* Psychiatric problems or unrealistic expectations
* Lack of opposing dentition in the area of interest
* Patients with poor root canal treatment
* Patients with parafunctional habits (eg. Bruxism)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Measuring number of Fracture | one year
  using USPHS criteria for clinical evaluation

SECONDARY OUTCOMES:
Degree of Marginal adaptation | one year
  using USPHS criteria for clinical evaluation
Degree of Marginal discoloration | one year
  using USPHS criteria for clinical evaluation
Presence of Caries | one year
  using USPHS criteria for clinical evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt